CLINICAL TRIAL: NCT00980486
Title: Effects of Maternal Obesity on Tissue Concentrations of Prophylactic Antibiotics During Cesarean Delivery
Brief Title: Obesity and Antibiotic Tissue Concentration
Status: Completed | Type: Observational
Sponsor: MemorialCare (Other)
Collaborators: University of California, Irvine (Other)
Responsible Party: Kenneth Chan MD, Long Beach Memorial Medical Center
Other Study IDs: 587-08
Record Dates: First submitted 2009-09-18; First posted 2009-09-21 (Estimated); Last update posted 2010-10-08 (Estimated); Status verified 2010-09

CONDITIONS: Obesity
Keywords: Antibiotic Concentration; Tissue; Obesity; Cesarean
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Adipose, myometrial and blood serum samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- BMI <30: BMI <30
- BMI 30-39: BMI 30-39
- BMI >40: BMI >40

SUMMARY:
The purpose of this study is to determine whether the dose of prophylactic antibiotics at the time of cesarean delivery requires adjustment in obese and overweight patients in order to achieve optimal antimicrobial activity.

DETAILED DESCRIPTION:
The majority of information regarding pharmacokinetics and pharmacodynamics (the action, properties and elimination of a drug in the body) of antibiotics is based on measurements of the serum and plasma concentrations. Current guidelines for surgical antibiotic prophylaxis have clearly demonstrated appropriate therapeutic levels within blood and serum levels, resulting in low incidence of postoperative bacteremia (bacteria in the blood) and sepsis (infection). Despite this, surgical site infections (SSI) remain the most common postoperative complication, affecting up to 20% of patients undergoing intra-abdominal surgery. Inadequate antibiotic penetration into the tissues of the surgical site, in spite of therapeutic serum levels, results in an environment that is susceptible to pathogens and subsequent infections. Antimicrobial tissue levels are influenced by volume of distribution, regional blood flow and biological properties of tissue. The ability of any drug to reach the tissue of interest is dictated by the relative amount of blood flow to that organ. While lungs and kidneys enjoy a robust blood supply, subcutaneous adipose tissue (fat) (the most frequent site of surgical site infections) receives a small fraction of the cardiac output. Obesity creates an increased volume of distribution, thereby resulting in a greater dilution of antibiotics when compared to non-obese subjects. Moreover, this change in volume of distribution is achieved primarily by increasing the relative amount of poorly perfused adipose tissue. Therefore, it should come as no surprise that obesity is a significant risk factor for surgical site infections.

The rate of obesity in the United States has shown a steady increase and more than doubled in the last twenty-five years from 15% in 1980 to 32.9% in 2004. Moreover, nearly one third of women of reproductive age are obese and approximately 6% are extremely obese. In addition to the usual health related concerns, obesity significantly increases the rate of complications associated with pregnancy. In particular, several studies have demonstrated an increased incidence of cesarean delivery associated to maternal obesity. Cesarean delivery rates, much like obesity rates, have witnessed a tremendous surge in the last few decades and now account for approximately 30% of all deliveries or nearly 1.2 million procedures. Surgical site infections associated with cesarean delivery include wound infections and endomyometritis (infection in the uterus), with rates ranging from 7% to 20% depending on the demographic and obstetric variables. Despite these alarming trends there is a paucity of data regarding antimicrobial activity of prophylactic antibiotics in tissues and the effects of maternal obesity on these concentrations at the time of cesarean delivery.

While the rates of cesarean deliveries have reached a plateau at around 30% in recent years, the rates of obesity continue to climb unabated. As the attributes of the population evolve over the course of time so must the guidelines and management adapt to the individuals in our care.

ELIGIBILITY:
Inclusion Criteria:

* Patients at term (> 37 weeks) undergoing a cesarean delivery.

Exclusion Criteria:

* Women younger than 18 years,
* Pre-gestational diabetes,
* Chronic hypertension,
* Collagen vascular disease,
* Multiple gestation,
* Contraindications to cefazolin administration (known anaphylactic reaction to penicillins or known cephalosporin allergy),
* Any exposure to cephalosporins in one week prior to cesarean section, OR
* Need for emergent cesarean delivery or diagnosis of chorioamnionitis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients requiring cesarean delivery under non-emergent circumstances
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2009-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To assess the effects of maternal obesity on the concentrations and adequacy of antimicrobial activity of prophylactically administered antibiotics within tissues (subcutaneous adipose and myometrial) at the time of cesarean delivery. | 6 weeks

SECONDARY OUTCOMES:
To assess the concentrations and adequacy of antimicrobial activity of prophylactically administered antibiotics within tissues (subcutaneous adipose and myometrial) at the time of cesarean delivery. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Chan, MD, Principal Investigator — Long Beach Memorial Medical Center
Locations (2):
- United States (2):
  - Women's Pavilion at Miller Children's Hospital, Long Beach, California
  - University of California Irvine Medical Center, Orange, California

REFERENCES:
- [Derived] Pevzner L, Swank M, Krepel C, Wing DA, Chan K, Edmiston CE Jr. Effects of maternal obesity on tissue concentrations of prophylactic cefazolin during cesarean delivery. Obstet Gynecol. 2011 Apr;117(4):877-882. doi: 10.1097/AOG.0b013e31820b95e4. PMID 21422859